CLINICAL TRIAL: NCT06785012
Title: A Randomized, Double-blind, Multicenter, Placebo-controlled, Proof-of-Concept Study to Evaluate the Efficacy, Safety, and Tolerability of JNJ-89495120 as Monotherapy in Adult Participants With Major Depressive Disorder (MDD)
Brief Title: A Study to Explore the Efficacy of JNJ-89495120 in the Treatment of Major Depressive Disorder
Acronym: Moonlight-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 89495120MDD2001; 89495120MDD2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-01-15; First posted 2025-01-20 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: JNJ-89495120 Dose A (Experimental): Participants will receive JNJ-89495120 dose A during the double-blind (DB) treatment phase in Period 1 and Period 2 of the study.
  Interventions: Drug: JNJ-89495120
- Arm 2: JNJ-89495120 Dose A and Dose B (Experimental): Participants will receive JNJ-89495120 dose A in Period 1 followed by JNJ-89495120 dose B in Period 2 during the DB treatment phase of the study.
  Interventions: Drug: JNJ-89495120
- Arm 3: Placebo Group (Placebo Comparator): Participants will receive placebo matched to JNJ-89495120 during the DB treatment phase in Period 1 and Period 2 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-89495120 — JNJ-89495120 will be administered.
  Arms: Arm 1: JNJ-89495120 Dose A; Arm 2: JNJ-89495120 Dose A and Dose B
Drug: Placebo — Placebo will be administered.
  Arms: Arm 3: Placebo Group

SUMMARY:
The purpose of this study is to evaluate how well JNJ-89495120 works (anti-depressant effects) and how well it is tolerated as compared to placebo on reducing the symptoms of depression in participants with major depressive disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* Primary psychiatric diagnosis of recurrent major depressive disorder, without psychotic features, based on clinical assessment using diagnostic and statistical manual of mental disorders (DSM)-5 criteria and confirmed with the mini international neuropsychiatric interview (MINI)
* Participant had to have at least one previous major depressive disorder (MDD) episode prior to their current episode
* Were first diagnosed with depression before the age of 55
* Are in a current episode of depression: Episode length must be at least 2 months but not longer than 24 months
* Have taken 0, 1, or 2 treatments for depression in your current episode
* Body mass index (BMI) within the range 18 to 35 kilograms per square meter (kg/m^2) at screening

Exclusion Criteria:

* Treatment with vagus nerve stimulation (VNS), electroconvulsive therapy (ECT), transcranial magnetic stimulation (TMS), deep brain stimulation (DBS), or ketamine/esketamine within the current or past major depressive episodes
* Current or past DSM-5 diagnosis of bipolar disorder, psychotic disorders, borderline personality disorder, antisocial personality disorder, or current obsessive-compulsive disorder
* Post-traumatic stress disorder within the past three years of screening
* Dementia, any dementing disease, intellectual disability, or neurocognitive disorder
* History of Alcohol and Substance use disorders within 6 months of screening, with the exclusion of nicotine, caffeine, and mild cannabis use disorder, according to the MINI and Clinical Assessment
* Known allergies, hypersensitivity, or intolerance to JNJ-89495120 or its excipients

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-12-26 (Actual); Primary Completion 2026-06-26 (Estimated); Study Completion 2026-06-26 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score to Day 5 | Baseline up to Day 5
  The MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.

SECONDARY OUTCOMES:
Change from Baseline in MADRS Total Score to Day 2 | Baseline up to Day 2
  The MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition.
Change from Baseline in Clinician Global Impression-Severity (CGI-S) Scale Score to Days 2 and 5 | Baseline up to Day 2 and Day 5
  The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness. The CGI-S evaluates the severity of psychopathology on a scale of 1 to 7. Participant is assessed on severity of illness at the time of rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. Higher score indicating greater severity.
Change from Baseline in Symptoms of Major Depressive Disorder Scale (SMDDS) Total Score to Day 5 | Baseline up to Day 5
  The SMDDS is a 16-item patient reported outcome (PRO) measure. Each item is rated by the participant according to a 5-point Likert scale, where 0 denotes "Not at all" or "Never" and 4 denotes "Extremely" or "Always". Before summing the items to create a total score, item 11 and item 12 are combined into a single score by selecting the highest severity on either item. The total score is then created by summing the responses on the 15 items, which range from 0 to 60. Higher score indicates more severe depressive symptomatology.
Change from Baseline in Generalized Anxiety Disorder-7 (GAD-7) Scale Score to Day 5 | Baseline up to Day 5
  The GAD-7 scale is a self-administered questionnaire designed to measure anxiety. GAD-7 has seven items, which measure frequency of various signs of GAD using a 4-point Likert scale (where, Not at all = 0, Several days = 1, More than half the days = 2, and Nearly every day = 3). The total score ranges from 0 to 21 with increasing scores indicative of greater severity of symptoms of anxiety. Severity of anxiety on the GAD-7 is rated as follows: none (0-4), mild (5-9), moderate (10-14) and severe (15-21).
Number of Participants with Adverse Events (AEs) | Up to approximately 18 weeks
  An AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Number of Participants with Abnormalities in Vital Signs Parameters | Up to approximately 18 weeks
  Participants with abnormalities in vital signs (supine blood pressure, pulse/heart rate, respiratory rate, oral temperature) parameters will be reported.
Number of Participants with 12-Lead Electrocardiogram (ECG) Abnormalities | Up to approximately 18 weeks
  Participants with 12-lead ECG abnormalities will be reported.
Number of Participants With Abnormalities in Laboratory Parameters | Up to approximately 18 weeks
  Participants with abnormalities in clinical laboratory parameters (hematology and serum chemistry) will be reported.
Number of Participants Reporting Changes in Weight/Body Mass Index (BMI) | Up to approximately 18 weeks
  Participants with changes in weight/BMI will be reported.
Suicidal Ideation Assessment Using Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to approximately 18 weeks
  The C-SSRS scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 'yes/no' items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Only items with yes responses are listed. Worsening of suicidal ideation was an increase in severity of suicidal ideation from baseline.
Change from Baseline in Cognitive Functioning Measured by the Hopkins Verbal Learning Test-Revised (HVLT-R) | From Baseline up to 4 weeks
  The HVLT-R, a measure of verbal learning and memory, is a 12-item word list recall test. Administration includes 3 learning trials, a delayed recall (20-minute) trial, and a 24-word recognition list (including 12 target and 12 foil words). The test administrator reads instructions and word lists aloud, and records words recalled/recognized by the participant. Three learning trials are combined to calculate a total recall score learning, delayed recall, and recognition trials.
Change from Baseline in Cognitive Functioning Measured by the Digit Symbol Substitution Test (DSST) | From Baseline up to 4 weeks
  The DSST is recognized as covering all of the cognitive performance aspects: speed of processing, executive functioning, and attention. The DSST measures attention, working memory, sustained visual attention and psychomotor speed. Participants are given a table that pairs digits and symbols, and asked to decipher a code using the table, completing as many as possible in 90 seconds.
Plasma Concentrations of JNJ-89495120 | Pre-dose (0 hours), and Post-dose on Days 1, 5 and 13
  Plasma concentrations of JNJ-89495120 will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (41):
- United States (41):
  - UAB Huntsville Regional Medical Campus, Huntsville, Alabama
  - Chandler Clinical Trials, Chandler, Arizona
  - IMA Clinical Research PC, Phoenix, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - CI Trials, Bellflower, California
  - Wake Research PRI Encino, Encino, California
  - National Institute Of Clinical Research, Garden Grove, California
  - WR-Newport Beach, Newport Beach, California
  - ATP Clinical Research, Orange, California
  - Anderson Clinical Research, Redlands, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Lumos Clinical Research Center LLC, San Jose, California
  - Syrentis Clinical Research, Santa Ana, California
  - Viking Clinical Research Ltd, Temecula, California
  - Sunwise Clinical Research, Walnut Creek, California
  - Mountain View Clinical Research, Denver, Colorado
  - Gulfcoast Medical Research Center, Fort Myers, Florida
  - The Medici Medical Research, Hollywood, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - K2 Medical Research, Maitland, Florida
  - Pharmax Research Clinic Inc, Miami, Florida
  - Wellness Research Center, Miami, Florida
  - Best Choice Medical and Research Service, Pembroke Pines, Florida
  - Interventional Psychiatry of Tampa Bay, Tampa, Florida
  - Synexus Clinical Research US Inc, Atlanta, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Indiana University IU Health, Indianapolis, Indiana
  - DelRicht Research, New Orleans, Louisiana
  - CBH Health, Gaithersburg, Maryland
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Integrative Clinical Trials LLC, Brooklyn, New York
  - Patient Priority Clinical Sites LLC, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - OSU Department of Psychiatry and Behavioral Health, Columbus, Ohio
  - Paradigm Research Professionals, LLC, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Revival Research Institute LLC, Sherman, Texas
  - Alpine Research Organization, Clinton, Utah
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency